CLINICAL TRIAL: NCT02798354
Title: Reducing Diagnostic Errors in Primary Care Pediatrics
Brief Title: Reducing Diagnostic Errors in Primary Care Pediatrics (Project RedDE)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: American Academy of Pediatrics (Other)
Responsible Party: Principal Investigator, Michael Rinke, Associate Professor, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2014-3980
Record Dates: First submitted 2016-05-25; First posted 2016-06-14 (Estimated); Results first posted 2019-12-16 (Actual); Last update posted 2019-12-16 (Actual); Status verified 2019-12

CONDITIONS: Diagnostic Errors
Keywords: Depression; Blood Pressure; Anemias, Iron-Deficiency; Streptococcal Infections; Sexually Transmitted Diseases; Lead Poisoning, Nervous System, Childhood; Thyrotropin
MeSH Terms: conditions — Depression; Anemia, Iron-Deficiency; Streptococcal Infections; Sexually Transmitted Diseases; Lead Poisoning, Nervous System, Childhood

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Reduce Elevated Blood Pressure Errors First (Experimental): Will provide baseline data on elevated blood pressure diagnosis and first intervene to reduce missed opportunities for elevated blood pressure diagnosis. Will then intervene to reduce missed opportunities for depression diagnosis and finally, intervene to reduce delayed diagnosis attributable to abnormal laboratory values.
  Quality Improvement Collaborative Intervention will consist of behavioral components, i.e., training, interactions with experts, root cause analyses of errors, idea sharing, best practices dissemination, etc.
  Interventions: Behavioral: Quality Improvement Collaborative
- Reduce Depression Errors First (Experimental): Will provide baseline data on depression diagnosis and first intervene to reduce missed opportunities for depression diagnosis. Will then intervene to reduce delayed diagnosis attributable to abnormal laboratory values and finally, intervene to reduce missed opportunities for elevated blood pressure diagnosis.
  Quality Improvement Collaborative Intervention will consist of behavioral components, i.e., training, interactions with experts, root cause analyses of errors, idea sharing, best practices dissemination, etc.
  Interventions: Behavioral: Quality Improvement Collaborative
- Reduce Lab Related Errors First (Experimental): Will provide baseline data on delayed diagnosis attributable to abnormal laboratory values and first intervene to reduce delayed diagnosis attributable to abnormal laboratory values. Will then intervene to reduce missed opportunities for elevated blood pressure diagnosis results and finally, to reduce missed opportunities for depression diagnosis.
  Quality Improvement Collaborative Intervention will consist of behavioral components, i.e., training, interactions with experts, root cause analyses of errors, idea sharing, best practices dissemination, etc.
  Interventions: Behavioral: Quality Improvement Collaborative

INTERVENTIONS:
Behavioral: Quality Improvement Collaborative — 1)Every 8 month 1-2 day interactive webinar learning sessions 2)Monthly webinars sharing best practices 3)Monthly team interactions with dedicated QI coach 4)Monthly data submission on both process and outcome measures 5)Monthly data feedback both at aggregate level with full inter-team transparency as well as at institutional level 6)Monthly mini root cause analyses performed on 1 error at each site 7)Multidisciplinary teams consisting of at least a physician, nurse, and office practice associate 8)Instruction on best practices from content area experts in QI, diagnostic errors, hypertension, mental health, leadership, behavior change, Model for Understanding Success in Quality (MUSIQ) and EHRs 9)Ongoing sharing of best ideas and barriers/issues among institutional teams

SUMMARY:
The proposal will focus on 3 specific, high-risk, pediatric ambulatory diagnostic errors each representing a unique dimension of diagnostic assessment: evaluation of symptoms, evaluation of signs and follow-up of diagnostic tests. Adolescent depression (i.e. symptoms) affects nearly 10% of teenagers, is misdiagnosed in almost 75% of adolescents and causes significant morbidity. Pediatric elevated blood pressure (signs) is misdiagnosed in 74-87% of patients, often due to inaccurate application of blood pressure parameters that change based on age, gender and height. Actionable pediatric laboratory values (diagnostic tests) are potentially delayed up to 26% of the time in preliminary investigations and 7-65% in adults, leading to harm and malpractice claims.

The investigators propose to conduct a multisite, prospective, stepped wedge cluster randomized trial testing a quality improvement collaborative (QIC) intervention within the American Academy of Pediatrics' Quality Improvement Innovation Networks (QuIIN) to reduce the incidence of pediatric primary care diagnostic errors. QuIIN is a national network of over 300 primary care practices, ranging from tertiary care academic medical centers to single practitioner private practices, interested in and experienced with QICs. Because many processes are likely to be common across diagnostic errors in outpatient settings, a multifaceted intervention, such as a QIC, has a high likelihood of success and broad applicability across populations. Preparatory inquiries to QuIIN primary care providers suggest high interest in reducing these 3 diagnostic errors and provider agreement with randomization to evaluate diagnostic error interventions. Practices will be randomized to one of three groups, with each group collecting retrospective baseline data on one error above, and then intervening to reduce that error during the first eight months. Each group will concurrently collect control data on an error they are not intervening on during those eight months. Following those eight months, the groups will continue intervening on their first error, begin intervening on the error they were a control site for, and begin collecting data on the third error for which they will be a control site for. Finally, in the final eight months, all groups will intervene on all three errors. A second wave of practices will be recruited to join the groups after eight months and will only intervene on two of the three errors.

DETAILED DESCRIPTION:
Objectives:

Primary

• To determine whether a QIC consisting of evidence-based best-practice methodologies, mini-root cause analyses, data sharing, and behavior change techniques, is associated with a reduction in 3 specific diagnostic error rates in a national group of pediatric primary care practices.

* Hypothesis 1: Implementation of a QIC will lead to a 40% reduction in missed diagnosis of adolescent depression.
* Hypothesis 2: Implementation of a QIC will lead to a 30% reduction in missed diagnosis of pediatric elevated blood pressure.
* Hypothesis 3: Implementation of a QIC will lead to a 45% reduction in delayed diagnosis of actionable laboratory results.

Secondary

* To determine if a QIC's effect changes for wave 1 versus wave 2 participants, or for the second versus the first error a practice intervenes on.
* To further investigate the epidemiology of three ambulatory pediatric diagnostic errors: missed diagnosis of adolescent depression, missed diagnosis of pediatric elevated blood pressure, and delayed diagnosis of actionable laboratory results.
* To evaluate patient outcomes related to these diagnoses including outcomes after positive depression screening, missed elevated blood pressure screening and delayed diagnosis of actionable laboratory values.

ELIGIBILITY:
Inclusion Criteria:

* The investigators will include 30 primary care pediatric practices that are part of the American Academy of Pediatrics' QuIIN (Quality Improvement Innovation Networks) organization. The second wave will recruit 15 additional practices.
* Practices must have sufficient volumes of adolescent well child visits (17 per month) and all well child visits (30 per month), and be able to query their EHR systems in order to be included in the study

Min Age: 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13853 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2017-10-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- American Academy of Pediatrics, Elk Grove Village, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bundy DG, Singh H, Stein RE, Brady TM, Lehmann CU, Heo M, O'Donnell HC, Rice-Conboy E, Rinke ML. The design and conduct of Project RedDE: A cluster-randomized trial to reduce diagnostic errors in pediatric primary care. Clin Trials. 2019 Apr;16(2):154-164. doi: 10.1177/1740774518820522. Epub 2019 Feb 5. PMID 30720339

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of note, initial control data were collected prior to the first Intervention Period
Units Other Than Participants: Clinics
Groups:
- Group 1: Blood Pressure, Depresion, Labs; Group 2: Depression, Labs, Blood Pressure; Group 3: Labs, Blood Pressure, Depression: A national cohort of pediatric practices enrolled in a Quality Improvement Collaborative intervention focused on reducing three errors of interest: blood pressure, labs and depression diagnoses. Each practice was cluster-randomized to collect control data on and then start working to reduce one of the three errors. During this first nine-month action phase, they also collected control data on a second error. Subsequently, practices worked to reduce this second error during an eight month action phase, while collecting control data on a third error. Finally, they worked to reduce this third error. During the second and third phases, they continued to collect data on the first and second errors.
Period: First Intervention Period
Arm/Group | Group 1: Blood Pressure, Depresion, Labs | Group 2: Depression, Labs, Blood Pressure | Group 3: Labs, Blood Pressure, Depression
Started (Clinic attrition occurred after enrollment due to data collection burden) | 1184; 14 Clinics | 2176; 16 Clinics | 990; 13 Clinics
Control Data Error 1 | 440; 11 Clinics | 549; 10 Clinics | 345; 10 Clinics
Intervention Data Error 1 | 744; 11 Clinics | 1627; 10 Clinics | 645; 10 Clinics
Completed | 1184; 11 Clinics | 2176; 10 Clinics | 990; 10 Clinics
Not Completed | 0; 3 Clinics | 0; 6 Clinics | 0; 3 Clinics
Period: Second Intervention Period
Arm/Group | Group 1: Blood Pressure, Depresion, Labs | Group 2: Depression, Labs, Blood Pressure | Group 3: Labs, Blood Pressure, Depression
Started | 2617; 11 Clinics | 1047; 10 Clinics | 1368; 10 Clinics
Control Data Error 2 | 1378; 11 Clinics | 593; 10 Clinics | 668; 9 Clinics
Intervention Data Error 2 | 1239; 11 Clinics | 454; 9 Clinics | 700; 10 Clinics
Completed | 2617; 11 Clinics | 1047; 9 Clinics | 1368; 10 Clinics
Not Completed | 0; 0 Clinics | 0; 1 Clinics | 0; 0 Clinics
Period: Third Intervention Period
Arm/Group | Group 1: Blood Pressure, Depresion, Labs | Group 2: Depression, Labs, Blood Pressure | Group 3: Labs, Blood Pressure, Depression
Started | 746; 11 Clinics | 1010; 9 Clinics | 2715; 10 Clinics
Control Data Error 3 | 419; 11 Clinics | 620; 9 Clinics | 1467; 10 Clinics
Intervention Data Error 3 | 327; 11 Clinics | 390; 9 Clinics | 1248; 10 Clinics
Completed | 746; 11 Clinics | 1010; 9 Clinics | 2715; 10 Clinics
Not Completed | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics

BASELINE CHARACTERISTICS:
Population: Each error had variable numbers of patients in the intervention and control groups
Groups:
- Reduce Elevated Blood Pressure Errors; Reduce Depression Errors; Reduce Lab Related Errors: A national cohort of pediatric practices enrolled in a Quality Improvement Collaborative intervention focused on reducing three errors of interest: blood pressure, labs and depression diagnoses. Each practice was cluster-randomized to collect control data on and then start working to reduce one of the three errors. During this first nine-month action phase, they also collected control data on a second error. Subsequently, practices worked to reduce this second error during an eight month action phase, while collecting control data on a third error. Finally, they worked to reduce this third error. During the second and third phases, they continued to collect data on the first and second errors. Data presented aggregates all control and intervention phase data respectively, from all three cohorts.
- Total: Total of all reporting groups
Arm/Group | Reduce Elevated Blood Pressure Errors | Reduce Depression Errors | Reduce Lab Related Errors | Total
Number analyzed (Participants) | 3562 | 7508 | 2783 | 13853
Age, Categorical [Count of Participants; unit: Participants] — Population: Each error had an intervention and control group
  Participants
    Intervention Group: number analyzed (Participants) | 1834 | 4114 | 1426 | 7374
    Intervention Group: <=18 years | 1805 | 3967 | 1332 | 7104
    Intervention Group: Between 18 and 65 years | 29 | 147 | 94 | 270
    Intervention Group: >=65 years | 0 | 0 | 0 | 0
    Control Group: number analyzed (Participants) | 1728 | 3394 | 1357 | 6479
    Control Group: <=18 years | 1695 | 3277 | 1282 | 6254
    Control Group: Between 18 and 65 years | 33 | 117 | 75 | 225
    Control Group: >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Each error had an intervention and control group
  Participants
    Intervention Group: number analyzed (Participants) | 1834 | 4114 | 1426 | 7374
    Intervention Group: Female | 880 | 2094 | 742 | 3716
    Intervention Group: Male | 954 | 2020 | 684 | 3658
    Control Group: number analyzed (Participants) | 1728 | 3394 | 1357 | 6479
    Control Group: Female | 836 | 1677 | 693 | 3206
    Control Group: Male | 892 | 1717 | 664 | 3273
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Insurance Status [Count of Participants; unit: Participants] — Population: Each error had an intervention and control group
  Participants
    Intervention Group: number analyzed (Participants) | 1834 | 4114 | 1426 | 7374
    Intervention Group: Private Insurance | 466 | 1086 | 322 | 1874
    Intervention Group: Non-private Insurance | 1368 | 3028 | 1104 | 5500
    Control Group: number analyzed (Participants) | 1728 | 3394 | 1357 | 6479
    Control Group: Private Insurance | 477 | 1011 | 322 | 1810
    Control Group: Non-private Insurance | 1251 | 2383 | 1035 | 4669

OUTCOME MEASURES:

1. Primary Outcome: Number of Adolescents Diagnosed With Depression Seen in Well Child Visits
Description: Patients >=11 years old with documentation of major depression or subsyndromal depression diagnoses in the medical record
Time Frame: Collected Monthly (5-9 baseline months and 8-9 intervention months depending on the enrolled cohort)
Measure: Count of Participants; unit: Participants
Groups:
- Control Group: Patients included at all practices during practices' depression control phase
- Intervention Group: Patients included at all practices during pratices' depression intervention phase
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 3394 | 4114
Participants | 233 | 443
Statistical Analysis 1: Comparison: Control Group vs Intervention Group; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Risk Difference (RD) = 3.9, 95% CI 2-sided [2.4 to 5.3] — Fitted by generalized mixed-effects model with potential clustering effects of practices and months taken into account; adjusted for age, sex, insurance, and wave

2. Primary Outcome: Number of Patients With Elevated Blood Pressure Measured and Appropriately Acted on by Providers
Description: Systolic or Diastolic Blood Pressure >= 90th percentile for age, gender and height or >=120/80 in >=3 years old patients at well child visits and at least one of: 1) provider repeated blood pressure, 2) clinic note mentions elevated blood pressure/hypertension 3) plan included recheck or evaluation of blood pressure, or 4) ordering laboratory or other studies to evaluate elevated blood pressure
Time Frame: Collected Monthly (5-9 baseline months and 8-9 intervention months depending on the enrolled cohort)
Measure: Count of Participants; unit: Participants
Groups:
- Control Group: Patients included at all practices during practices' BP control phase
- Intervention Group: Patients included at all practices during practices' BP intervention phase
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 1728 | 1834
Participants | 969 | 1378
Statistical Analysis 1: Comparison: Control Group vs Intervention Group; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Risk Difference (RD) = 16, 95% CI 2-sided [12.3 to 20] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Number of Patients With Abnormal Laboratory Results With Appropriate Actions Without Delay
Description: Documented action step for first positive within 30 days:
  1. Hemoglobin (Hgb) less than 11 and mean corpuscular volume (MCV) less than 75 in 1 or 2 year old without documentation of beginning iron, sending iron studies or family conversation
  2. Lead greater than 5 without documentation of family conversation on lead remediation or plan to retest
  Documented action step for first positive within 7 days:
  1. Positive Gonorrhea, Chlamydia, Syphilis or Human immunodeficiency virus (HIV) test without documentation of antibiotics begun or referral to HIV specialist
  2. Positive group A streptococcal throat culture with negative rapid group A streptococcal test without documentation of antibiotics begun or family conversation
  3. Thyroid stimulating hormone (TSH) less than 0.5 or greater than 4.5 in greater than 1 year old without plan to repeat lab values or referral to endocrinologist
Time Frame: Collected Monthly (5-9 baseline months and 8-9 intervention months depending on the enrolled cohort)
Measure: Count of Participants; unit: Participants
Groups:
- Control Group: Patients included at all practices during practices' Labs control phase
- Intervention Group: Patients included at all practices during practices' Labs intervention phase
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 1357 | 1426
Participants | 1273 | 1329
Statistical Analysis 1: Comparison: Control Group vs Intervention Group; Test type: Superiority; p = 0.302, Mixed Models Analysis; Risk Difference (RD) = 1.1, 95% CI 2-sided [-1.0 to 3.1] — Fitted by generalized mixed-effects model with potential clustering effects of practices and months taken into account; adjusted for age, sex, insurance, lab test sent, and wave

4. Secondary Outcome: Number of Adolescents With Mental Health Addressed During Their Well Child Visit
Description: Provider screened for mental health concerns either with standard screening tool or clinical judgement and documented mental health concerns or no mental health concerns.
Time Frame: Collected Monthly (5-9 baseline months and 8-9 intervention months depending on the enrolled cohort)
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 3394 | 4114
Participants | 1782 | 3075
Statistical Analysis 1: Comparison: Control Group vs Intervention Group; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Risk Difference (RD) = 26.6, 95% CI 2-sided [22.4 to 30.7] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Number of Patients With Elevated Blood Pressures Measured and Blood Pressure Percentiles Documented in the Chart
Description: Systolic or Diastolic Blood Pressure >= 90th percentile for age, gender and height or >=120/80 in >=3 years old patients at well child visits with blood pressure percentiles documented per the 4th Report.
Time Frame: Collected Monthly (5-0 baseline months and 8-9 intervention months depending on the enrolled cohort)
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 1728 | 1834
Participants | 1233 | 1681
Statistical Analysis 1: Comparison: Control Group vs Intervention Group; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Risk Difference (RD) = 20.1, 95% CI 2-sided [16.2 to 24.1] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Number of Patients With Elevated Blood Pressures Measured and Recognized by Provider
Description: Systolic or Diastolic Blood Pressure >= 90th percentile for age, gender and height or >=120/80 in >=3 years old patients at well child visits with provider documentation of abnormal blood pressure or appropriate action taken
Time Frame: Collected Monthly (5-9 baseline months and 8-9 intervention months depending on the enrolled cohort)
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 1728 | 1834
Participants | 1013 | 1394
Statistical Analysis 1: Comparison: Control Group vs Intervention Group; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Risk Difference (RD) = 14, 95% CI 2-sided [10.3 to 17.7] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Number of Patients With Abnormal Laboratory Results Received and Recognized by Provider
Description: Provider documentation of abnormal laboratory value, of appropriate diagnosis (e.g. iron deficiency anemia) or appropriate action taken without delay as defined above.
Time Frame: Collected Monthly (5-9 baseline months and 8-9 intervention months depending on the enrolled cohort)
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 1357 | 1426
Participants | 1292 | 1339
Statistical Analysis 1: Comparison: Control Group vs Intervention Group; Test type: Superiority; p = 0.922, Mixed Models Analysis; Risk Difference (RD) = 0.1, 95% CI 2-sided [-1.8 to 1.9] — [estimate comment as in outcome 3, analysis 1]

8. Other Pre Specified Outcome: Percent of Clinics Reaching Pre-Determined Threshold for Providers With Laboratory Results Unread/Unacknowledged in Their Electronic Health Record (EHR) Inbox for More Than 72 Hrs
Description: Clinics reported percent of EHR inboxes with laboratory results unread/unacknowledged in their electronic health record (EHR) inbox for more than 72 hrs each month. They reported whether this percentage was equal to or less than 10%, the pre-determined threshold. They only collected this process measure until they were compliant with the threshold for 2 consecutive months.
Time Frame: Collected at 4 months
Measure: Count of Units; unit: Clinics
Units Other Than Participants: Clinics
Arm/Group | Intervention Group
Number analyzed (Participants) | 1426
Number analyzed (Clinics) | 30
Clinics | 27

9. Other Pre Specified Outcome: Percent of Clinics Reaching Pre-determined Threshold for Children Greater Than or Equal to 3 Yrs Old Receiving Blood Pressure Measurements at Triage for Well Child Visits
Description: Clinics reported percent of well child visit charts with blood pressure measurements at triage done each month. They reported whether this percentage was equal to or greater than 90%, the pre-determined threshold. They only collected this process measure until they were compliant with the threshold for 2 consecutive months.
Time Frame: Collected until 2 months
Measure: Count of Units; unit: Clinics
Units Other Than Participants: Clinics
Arm/Group | Intervention Group
Number analyzed (Participants) | 1834
Number analyzed (Clinics) | 30
Clinics | 27

10. Other Pre Specified Outcome: Percent of Clinics Reaching Predetermined Threshold for Adolescents Screened for Depression With Patient Health Questionnaire-9 Modified (PHQ-9M) During Well Child Visits
Description: Clinics reported percent of adolescent well child visit charts with depression screening done each month. They reported whether this percentage was equal to or greater than 90%, the pre-determined threshold. They only collected this process measure until they were compliant with the threshold for 2 consecutive months.
Time Frame: Collected monthly for 8 months when practice is intervening on this topic
Measure: Count of Units; unit: Clinics
Units Other Than Participants: Clinics
Arm/Group | Intervention Group
Number analyzed (Participants) | 4114
Number analyzed (Clinics) | 31
Clinics
  Percent of Clinics meeting threshold at 5 months | 15
  Percent of Clinics meeting threshold at 8 months | 21

ADVERSE EVENTS:
Description: As this quality improvement research study was considered low risk, no adverse event data was collected.
Groups:
- Reduce Elevated Blood Pressure Errors: Will provide baseline data on elevated blood pressure diagnosis and first intervene to reduce missed opportunities for elevated blood pressure diagnosis. Will then intervene to reduce missed opportunities for depression diagnosis and finally, intervene to reduce delayed diagnosis attributable to abnormal laboratory values. Each group provides control data and intervention data on all 3 errors in different sequences. Three Wave 2 practices were recruited to increase power and they intervened on only 2 errors.
  Quality Improvement Collaborative: 1)Every 8 month 1-2 day interactive webinar learning sessions 2)Monthly webinars sharing best practices 3)Monthly team interactions with dedicated QI coach 4)Monthly data submission on both process and outcome measures 5)Monthly data feedback both at aggregate level with full inter-team transparency as well as at institutional level 6)Monthly mini root cause analyses performed on 1 error at each site 7)Multidisciplinar
- Reduce Depression Errors: Will provide baseline data on depression diagnosis and first intervene to reduce missed opportunities for depression diagnosis. Will then intervene to reduce delayed diagnosis attributable to abnormal laboratory values and finally, intervene to reduce missed opportunities for elevated blood pressure diagnosis.
  Each group provides control data and intervention data on all 3 errors in different sequences. Two Wave 2 practices were recruited to increase power and they intervened on only 2 errors.
  Quality Improvement Collaborative: 1)Every 8 month 1-2 day interactive webinar learning sessions 2)Monthly webinars sharing best practices 3)Monthly team interactions with dedicated QI coach 4)Monthly data submission on both process and outcome measures 5)Monthly data feedback both at aggregate level with full inter-team transparency as well as at institutional level 6)Monthly mini root cause analyses performed on 1 error at each site 7)Multidisciplinary teams cons
- Reduce Lab Related Errors: Will provide baseline data on delayed diagnosis attributable to abnormal laboratory values and first intervene to reduce delayed diagnosis attributable to abnormal laboratory values. Will then intervene to reduce missed opportunities for elevated blood pressure diagnosis results and finally, to reduce missed opportunities for depression diagnosis. Each group provides control data and intervention data on all 3 errors in different sequences. Four Wave 2 practices were recruited to increase power and they intervened on only 2 errors.
  Quality Improvement Collaborative: 1)Every 8 month 1-2 day interactive webinar learning sessions 2)Monthly webinars sharing best practices 3)Monthly team interactions with dedicated QI coach 4)Monthly data submission on both process and outcome measures 5)Monthly data feedback both at aggregate level with full inter-team transparency as well as at institutional level 6)Monthly mini root cause analyses performed on 1 error at ea
Arm/Group | Reduce Elevated Blood Pressure Errors | Reduce Depression Errors | Reduce Lab Related Errors
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Practices enrolled in a QIC are likely not representative of all practices. Appropriate actions broadly defined. No direct chart review verifications. No data on 11 practices who left the study. Quasi-random chart review strategy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-21): https://cdn.clinicaltrials.gov/large-docs/54/NCT02798354/Prot_SAP_000.pdf